CLINICAL TRIAL: NCT04920448
Title: TOLERANCE STUDY OF N-ACETYLCYSTEINE FOR THROMBOLYSIS IN THE ACUTE PHASE OF ISCHEMIC STROKE / ETUDE DE TOLERANCE DE LA N-ACETYLCYSTEINE POUR LA THROMBOLYSE A LA PHASE AIGUË DE L'INFARCTUS CEREBRAL
Brief Title: N-ACETYLCYSTEINE FOR THROMBOLYSIS IN ACUTE STROKE
Acronym: NAC-S
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of patients
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-079
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Ischemic
Keywords: Thrombolysis; Hemorrhagic transformation; Alteplase; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- N-Acetylcysteine 150 mg/kg (Experimental): Single intravenous injection of N-Acetylcysteine (150 mg/kg in 15 minutes).
  Interventions: Drug: N-Acetyl cysteine

INTERVENTIONS:
Drug: N-Acetyl cysteine — Administered as specified in the treatment arm
  Other Names: HIDONAC

SUMMARY:
The primary objective of the study is to assess the safety of N-Acetylcysteine as a thrombolytic agent in acute ischemic stroke, especially regarding the risk of hemorrhagic transformation.

DETAILED DESCRIPTION:
Preclinical studies demonstrated that N-Acetylcysteine (NAC) is able to break von Willebrand Factor (VWF) multimers by bisulfide bond reduction. Since thrombi in stroke patients are rich in VWF, NAC could be used as a thrombolytic agent during the acute phase. This study aims at assessing the safety of NAC in combination with alteplase (rt-PA) at the acute phase of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with an acute ischemic stroke (non lacunar) as assessed by cerebral imaging (either CT or MRI), with or without visible vessel occlusion.
* Patient eligible to intravenous thrombolysis according to current criteria, including patients who will also benefit from endovascular treatment (if eligible).
* Personal or familial consent to participate in the study.

Exclusion Criteria:

* Known hypersensitivity to N-Acetylcysteine or to any excipient from the formulation.
* Coma and/or NIHSS <4 or ≥20.
* Daily treatment with Nitrovasodilator before the inclusion.
* Known asthma or chronic obstructive pulmonary disease requiring bronchodilatators or steroids.
* Participation to another interventional study if it requires administration of an experimental treatment in the first 3 days after NAC treatment.
* Women of childbearing age (age < or = to 50)
* Known history of prior treatment with vitamin-K antagonist or direct oral anticoagulant.
* Known history of severe hepatopathy including cirrhosis, portal hypertension (esophageal varices) and evolutive hepatopathy.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Symptomatic intracranial hemorrhagic transformation | 22 to 36 hours after treatment
  Rate of symptomatic hemorrhagic transformation according to the SITS-MOST criteria: a local or remote parenchymal hemorrhage on imaging 22 to 36 hours after treatment or earlier if the imaging scan was performed due to clinical deterioration combined with a neurological deterioration of >4 NIHSS points from baseline or from the lowest NIHSS score between baseline and 24 hours or leading to death within 24 hours.

SECONDARY OUTCOMES:
Extracranial hemorrhagic events | Up to 3 months after treatment
  Rate of extracranial hemorrhagic events
Treatment related side effects | Up to 3 months after treatment
  Rate of any drug related side effects according to the Common Terminology Criteria of Adverse Event 5.0.
Mortality and functional independence | 3 months after treatment
  Rate of mortality and functional independence at 3 months according to the modified Rankin scale (mRs)
Early neurological improvement | 24 hours after treatment
  Rate of early neurological improvement defined as an improvement of >4 NIHSS points 24 hours after treatment.
Plasma VWF multimers | Before, at 3 hours and at 24 hours after treatment
  Mean size of VWF multimers before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, Normandy, France

REFERENCES:
- [Background] Martinez de Lizarrondo S, Gakuba C, Herbig BA, Repesse Y, Ali C, Denis CV, Lenting PJ, Touze E, Diamond SL, Vivien D, Gauberti M. Potent Thrombolytic Effect of N-Acetylcysteine on Arterial Thrombi. Circulation. 2017 Aug 15;136(7):646-660. doi: 10.1161/CIRCULATIONAHA.117.027290. Epub 2017 May 9. PMID 28487393